CLINICAL TRIAL: NCT00346242
Title: Evaluation of Efficacy of Zoledronic Acid in Patients With Haemoglobin Syndromes (Thalassemia and Sicle Cell Anaemia) and Risk of Skeletal Events
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CZOL446EGR05
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Thalassemia
Keywords: thalassemia; zoledronic acid; skeletal events
MeSH Terms: conditions — Thalassemia | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid

SUMMARY:
The evaluation of efficacy is performed by laboratory monitoring of bone density and resorption markers and clinical monitoring of bone density improvement. This is a prospective, randomized, parallel group, single blind study of one year treatment with zoledronic acid every 6 months as compared to one year treatment with zoledronic acid every 3 months and to placebo every 3 months in patients with hemoglobin syndromes and risk of skeletal complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thalassaemia or sickle cell anaemia and bone density, z-scores < -1.5, in at least one of the examined sites
* Normal renal function. Urea and creatinine should not exceed > 2-fold the upper limit of normal (< 2 x ULN).

Exclusion Criteria:

-

Other protocol-defined inclusion / exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-03; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Bone density by means of bone densitometry with dual energy x-ray absorptiometry (DEXA) at three body sites (lumbar region, femoral head, wrist) prior to treatment initiation the start and at the end of treatment
N-telopeptide of type I collagen (NTx) levels, TRACP-5b, with ELISA, prior to the start of treatment initiation and every 3 or 6 months
Serum Bone alkaline phosphatase, Osteocalcin, OPG and S-RANKL with ELISA, prior to the start of treatment initiation, and every 3 or 6 months

SECONDARY OUTCOMES:
Biochemistry (Ca, P, urea/creatinine, SGOT/SGPT, ALT, γGT), endocrine and cardiac test prior to the start of treatment initiation and at 6 and 12 month.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Novartis Investigative Site, Athens, Greece

REFERENCES:
- [Derived] Voskaridou E, Christoulas D, Xirakia C, Varvagiannis K, Boutsikas G, Bilalis A, Kastritis E, Papatheodorou A, Terpos E. Serum Dickkopf-1 is increased and correlates with reduced bone mineral density in patients with thalassemia-induced osteoporosis. Reduction post-zoledronic acid administration. Haematologica. 2009 May;94(5):725-8. doi: 10.3324/haema-tol.2008.000893. PMID 19407319